CLINICAL TRIAL: NCT04070976
Title: Phase II Randomized Controlled Trial of Concomitant Chemoradiotherapy With Standard Fractionation Compared to Hypofractionated Concomitant Chemoradiotherapy Followed by Brachytherapy, for Clinical Stage III Cervical Cancer Patients
Brief Title: Chemotherapy and Pelvic Hypofractionated Radiation Followed by Brachytherapy for Cervical Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Institute of Cancerología (Other Government)
Responsible Party: Principal Investigator, David Cantu, Chief of clinical trials department, National Institute of Cancerología
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 019/036/ICI
Record Dates: First submitted 2019-08-22; First posted 2019-08-28 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Cervical Cancer
Keywords: hypofractionated radiotherapy; Brachytherapy
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard treatment (Active Comparator): Cisplatin 40mg/m2 weekly and concomitant pelvic radiotherapy (45 Gray/25 fractions) followed by brachytherapy 28Gray at point A.
  Interventions: Radiation: Standard therapy
- Experimental treatment (Experimental): Cisplatin 40mg/m2 weekly and hypofractionated concomitant external radiotherapy (37,50 Gray/15 fractions) followed by brachytherapy 28 Gray at point A.
  Interventions: Radiation: Hypofractionated therapy

INTERVENTIONS:
Radiation: Hypofractionated therapy — All patients will be treated with an external beam of 37.5 Gray in 15 fractions (2.5 Gray / fraction). They will be treated once a day, 5 days a week. If photon energy 6 MV or 10 MV is used, the patient should be treated with a 4-field technique using the anterior/posterior field and 2 lateral fields. The specification of the dose is in terms of a dose to a point at or near the center of the target volume. For all field dispositions, the dose specification point is the common isocenter of all beams.
  Arms: Experimental treatment
Radiation: Standard therapy — All patients will be treated with external beam radiotherapy with 50 Gray in 25 fractions (1.8-2 Gray / fraction). They will be treated once a day, 5 days a week. If photon energy 6 MV or 10 MV is used, the patient should be treated with a 4-field technique using anterior/posterior fields and 2 lateral fields. The specification of the dose is in terms of a dose to a point at or near the center of the target volume. For all field dispositions, the dose specification point is the common isocenter of all beams.
  Arms: Standard treatment

SUMMARY:
The main goal of this trial is to assess the safety and response rate to concomitant chemotherapy and external hypofractionated radiotherapy followed by brachytherapy in patients with clinical stage III cervical cancer. The trial will take place in the National Cancer Institute (INCan). Patients will be randomized into two groups: chemotherapy with external standard fractionated radiotherapy (45 Gy in 25 fractions) followed by brachytherapy or chemotherapy with external hypofractionated radiotherapy (37.5 Gy in 15 fractions) followed by brachytherapy.

DETAILED DESCRIPTION:
The primary endpoint will be to assess the safety and efficacy to concomitant chemoradiotherapy followed by brachytherapy in cervical cancer clinical stage III. Secondary endpoints comprises security profile, survival rates, quality of life and related costs.

The data obtained by this protocol will allow to determine the effect of hypofractionated radiation therapy and its possible adverse effects. Side effects will be classified according to version 4.03 of CTCAE guidelines. The highest CTCAE grade will be obtained for each type of event, for each patient and the Radiation Therapy Oncology Group (RTOG) scale will be applied to evaluate the events related to conventional and hypofractionated radiotherapy, as well as brachytherapy.

Quality of life (QOL) will be evaluated using EORTC QLQ-CX24 and EORTC QLQ-C30, both have been validated and available in Mexican Spanish.

Direct and indirect expenses related to the treatment will be evaluated based on the treatment costs stipulate by the institution and the information obtained by the social workers.

ELIGIBILITY:
Inclusion Criteria:

* Women over 18 years old
* Cervical Cancer at IIIA, IIIB y IIIC1 FIGO´s clinical stages
* Histology: squamous, adenosquamous or adenocarcinoma
* No previous treatment
* No distance metastases, discard by Positron Emission Tomography (PET)/CT
* Functional State ECOG (Eastern Cooperative Oncology Group) 0-2
* Complete Blood count obtained at least 14 days before admission to the study with adequate bone marrow function defined as:
* Absolute neutrophil count ≥ 1,500 cell/mm3
* Platelets ≥ 100,000 cell/mm3
* Hemoglobin ≥ 10.0 g/dl
* Leukocyte count ≥ 4000 cell/mm3
* Adequate Renal Function defined as:
* Serum Creatinine ≤ 1.5 mg/dl within 14 days before admission to the study
* Patients with HIV infection (human immunodeficiency virus) must have a CD4 cell count ≥ 350 cells / mm3 measured within 14 days prior to study entry (no HIV test is required)
* The patient must understand the protocol and provide the specific informed consent of the study before admission
* Negative pregnancy test

Exclusion Criteria:

* Patients who had chemotherapeutic, surgical and/or radiotherapy treatment for female reproductive tract pathologies
* Previous invasive neoplasia (except non-melanoma skin cancer) unless there is complete remission of the disease of 3 years minimum (For example, breast cancer or oral cavity cancer)
* Previous systemic chemotherapy for current cervical cancer, take into account that prior chemotherapy for a different cancer is accepted, as long as they have been at least 3 years
* Severe active or non-controlled co-morbidities, defined as:
* Unstable angina and/or congestive heart failure that required hospitalization in the last 6 months.
* Transmural myocardial infarction in the last 6 months.
* Acute bacterial or fungal infection requiring intravenous antibiotics at the beginning of the study.
* Chronic obstructive pulmonary disease exacerbation or another respiratory disease that requires hospitalization or that contraindicates the trial therapy at the time of admission.
* Crohn's disease or ulcerative colitis.
* Prior allergic reaction to cisplatin or other drugs based on platinum.
* Other factors that contraindicate experimental therapy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2024-07-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Acute and late toxicity | 2 years
  Number of Participants With Treatment-Related Adverse Events as Assessed by RTOG

SECONDARY OUTCOMES:
Treatment efficacy | 2 years
  Hypofractionated radiotherapy is similar in toxicity and disease control compared to standard external beam treatment
Disease-free survival rate | 2 years
  Number of participants dead of disease at two years according to kaplan-meyer analysis
Overall survival rate | 2 years
  Number ofpParticipants dead at two years according to kaplan-meyer analysis
Satisfaction assessed by EORTC | 2 years
  Assessed individual's overall satisfaction with life and general sense of personal well-being by ERTC QLQ-C30 and QLQ-CX24 questionaire
Direct and indirect costs related to treatment. | 2 years
  Direct costs related to the treatment. Indirect costs related to the treatment (transport, housing, food, etc.)

CONTACTS AND LOCATIONS:
Overall Officials: David F Cantú-deLeón, Principal Investigator — Instituto Nacional de Cancerologia de Mexico
Locations (1):
- David Cantu de Leon, Mexico City, Tlalpan, Mexico

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP
Time Frame: 2 years
Access Criteria: the data will be shared with scientific and academic institutions or research groups that study the same topic and with the regulatory and ethical authorities that require it, to ensure the quality and accuracy of the data.

REFERENCES:
- [Background] Ferlay J, Soerjomataram I, Dikshit R, Eser S, Mathers C, Rebelo M, Parkin DM, Forman D, Bray F. Cancer incidence and mortality worldwide: sources, methods and major patterns in GLOBOCAN 2012. Int J Cancer. 2015 Mar 1;136(5):E359-86. doi: 10.1002/ijc.29210. Epub 2014 Oct 9. PMID 25220842
- [Background] Gosvig CF, Huusom LD, Andersen KK, Duun-Henriksen AK, Frederiksen K, Iftner A, Svare E, Iftner T, Kjaer SK. Long-term follow-up of the risk for cervical intraepithelial neoplasia grade 2 or worse in HPV-negative women after conization. Int J Cancer. 2015 Dec 15;137(12):2927-33. doi: 10.1002/ijc.29673. Epub 2015 Jul 25. PMID 26139420
- [Background] Morris M, Eifel PJ, Lu J, Grigsby PW, Levenback C, Stevens RE, Rotman M, Gershenson DM, Mutch DG. Pelvic radiation with concurrent chemotherapy compared with pelvic and para-aortic radiation for high-risk cervical cancer. N Engl J Med. 1999 Apr 15;340(15):1137-43. doi: 10.1056/NEJM199904153401501. PMID 10202164
- [Background] Carlson RW, Scavone JL, Koh WJ, McClure JS, Greer BE, Kumar R, McMillian NR, Anderson BO. NCCN Framework for Resource Stratification: A Framework for Providing and Improving Global Quality Oncology Care. J Natl Compr Canc Netw. 2016 Aug;14(8):961-9. doi: 10.6004/jnccn.2016.0103. PMID 27496112
- [Background] Robin TP, Amini A, Schefter TE, Behbakht K, Fisher CM. Disparities in standard of care treatment and associated survival decrement in patients with locally advanced cervical cancer. Gynecol Oncol. 2016 Nov;143(2):319-325. doi: 10.1016/j.ygyno.2016.09.009. Epub 2016 Sep 16. PMID 27640961
- [Background] Greenup RA, Blitzblau RC, Houck KL, Sosa JA, Horton J, Peppercorn JM, Taghian AG, Smith BL, Hwang ES. Cost Implications of an Evidence-Based Approach to Radiation Treatment After Lumpectomy for Early-Stage Breast Cancer. J Oncol Pract. 2017 Apr;13(4):e283-e290. doi: 10.1200/JOP.2016.016683. Epub 2017 Mar 14. PMID 28291382
- [Background] Muckaden MA, Budrukkar AN, Tongaonkar HB, Dinshaw KA. Hypofractionated radiotherapy in carcinoma cervix IIIB: Tata Memorial Hospital experience. Indian J Cancer. 2002 Oct-Dec;39(4):127-34. PMID 12928570
- [Background] Zhang H, Wang JZ, Mayr N, Kong X, Yuan J, Gupta N, Lo S, Grecula J, Montebello J, Martin D, Yuh W. Fractionated grid therapy in treating cervical cancers: conventional fractionation or hypofractionation? Int J Radiat Oncol Biol Phys. 2008 Jan 1;70(1):280-8. doi: 10.1016/j.ijrobp.2007.08.024. Epub 2007 Oct 29. PMID 17967516
- [Background] Hoffman KE, Voong KR, Pugh TJ, Skinner H, Levy LB, Takiar V, Choi S, Du W, Frank SJ, Johnson J, Kanke J, Kudchadker RJ, Lee AK, Mahmood U, McGuire SE, Kuban DA. Risk of late toxicity in men receiving dose-escalated hypofractionated intensity modulated prostate radiation therapy: results from a randomized trial. Int J Radiat Oncol Biol Phys. 2014 Apr 1;88(5):1074-84. doi: 10.1016/j.ijrobp.2014.01.015. PMID 24661661
- [Background] Antoni S, Soerjomataram I, Moller B, Bray F, Ferlay J. An assessment of GLOBOCAN methods for deriving national estimates of cancer incidence. Bull World Health Organ. 2016 Mar 1;94(3):174-84. doi: 10.2471/BLT.15.164384. Epub 2016 Jan 28. PMID 26966328
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] Ferlay J, Colombet M, Soerjomataram I, Mathers C, Parkin DM, Pineros M, Znaor A, Bray F. Estimating the global cancer incidence and mortality in 2018: GLOBOCAN sources and methods. Int J Cancer. 2019 Apr 15;144(8):1941-1953. doi: 10.1002/ijc.31937. Epub 2018 Dec 6. PMID 30350310
- [Background] Bhatla N, Aoki D, Sharma DN, Sankaranarayanan R. Cancer of the cervix uteri. Int J Gynaecol Obstet. 2018 Oct;143 Suppl 2:22-36. doi: 10.1002/ijgo.12611. PMID 30306584
- [Background] FIGO Committee on Gynecologic Oncology. FIGO staging for carcinoma of the vulva, cervix, and corpus uteri. Int J Gynaecol Obstet. 2014 May;125(2):97-8. doi: 10.1016/j.ijgo.2014.02.003. Epub 2014 Feb 22. No abstract available. PMID 24630859
- [Background] Chuang LT, Temin S, Camacho R, Duenas-Gonzalez A, Feldman S, Gultekin M, Gupta V, Horton S, Jacob G, Kidd EA, Lishimpi K, Nakisige C, Nam JH, Ngan HYS, Small W, Thomas G, Berek JS. Management and Care of Women With Invasive Cervical Cancer: American Society of Clinical Oncology Resource-Stratified Clinical Practice Guideline. J Glob Oncol. 2016 May 25;2(5):311-340. doi: 10.1200/JGO.2016.003954. eCollection 2016 Oct. PMID 28717717
- [Background] Leath CA 3rd, Monk BJ. Twenty-first century cervical cancer management: A historical perspective of the gynecologic oncology group/NRG oncology over the past twenty years. Gynecol Oncol. 2018 Sep;150(3):391-397. doi: 10.1016/j.ygyno.2018.06.023. Epub 2018 Jun 27. PMID 29954593
- [Background] Kirwan JM, Symonds P, Green JA, Tierney J, Collingwood M, Williams CJ. A systematic review of acute and late toxicity of concomitant chemoradiation for cervical cancer. Radiother Oncol. 2003 Sep;68(3):217-26. doi: 10.1016/s0167-8140(03)00197-x. PMID 13129628
- [Background] Koh WJ, Abu-Rustum NR, Bean S, Bradley K, Campos SM, Cho KR, Chon HS, Chu C, Clark R, Cohn D, Crispens MA, Damast S, Dorigo O, Eifel PJ, Fisher CM, Frederick P, Gaffney DK, Han E, Huh WK, Lurain JR, Mariani A, Mutch D, Nagel C, Nekhlyudov L, Fader AN, Remmenga SW, Reynolds RK, Tillmanns T, Ueda S, Wyse E, Yashar CM, McMillian NR, Scavone JL. Cervical Cancer, Version 3.2019, NCCN Clinical Practice Guidelines in Oncology. J Natl Compr Canc Netw. 2019 Jan;17(1):64-84. doi: 10.6004/jnccn.2019.0001. PMID 30659131
- [Background] Das S, Subhashini J, Rami Reddy JK, KantiPal S, Isiah R, Oommen R. Low-dose fractionated radiation and chemotherapy prior to definitive chemoradiation in locally advanced carcinoma of the uterine cervix: Results of a prospective phase II clinical trial. Gynecol Oncol. 2015 Aug;138(2):292-8. doi: 10.1016/j.ygyno.2015.05.020. Epub 2015 May 23. PMID 26013695
- [Background] Duenas-Gonzalez A, Zarba JJ, Patel F, Alcedo JC, Beslija S, Casanova L, Pattaranutaporn P, Hameed S, Blair JM, Barraclough H, Orlando M. Phase III, open-label, randomized study comparing concurrent gemcitabine plus cisplatin and radiation followed by adjuvant gemcitabine and cisplatin versus concurrent cisplatin and radiation in patients with stage IIB to IVA carcinoma of the cervix. J Clin Oncol. 2011 May 1;29(13):1678-85. doi: 10.1200/JCO.2009.25.9663. Epub 2011 Mar 28. PMID 21444871
- See also: Human papillomavirus (HPV) and cervical cancer [Internet] — https://www.who.int/news-room/fact-sheets/detail/human-papillomavirus-(hpv)-and-cervical-cancer